CLINICAL TRIAL: NCT00763126
Title: The Effect of the Presence of a Spouse on the Parturient's and Her Spouse's Stress Level During Epidural Analgesia During Labor as Measured by Salivary Amylase
Brief Title: Does Having a Spouse Present During Epidural Analgesia Affect Stress Levels in the Parturient and Her Spouse?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sharon Orbach-Zinger, M.D, Anesthesiology department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5053
Record Dates: First submitted 2008-09-28; First posted 2008-09-30 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Labor Pain
Keywords: parturient; epidural analgesia; labor; spouse; Stress levels; Salivary amylase
MeSH Terms: conditions — Labor Pain

ARMS (2):
- Spouse present, (Active Comparator)
  Interventions: Behavioral: stress level
- spouse absent (Active Comparator)
  Interventions: Behavioral: stress level

INTERVENTIONS:
Behavioral: stress level — Stress levels

SUMMARY:
It is unclear the effect of a spouse's presence on the partureint's and the spouse's stress level during the performance of epidural analgesia during labor.

Couples will be randomized to two groups: one group where the spouse is present during the performance of epidural analgesia and the second where the spouse is not present.

Before and after epidural anlgesia, both the spouse and parturient will be have their blood pressure and pulse checked. In addition, both will have their salivary amylase measured.

Salivary amylase is an enzyme whic has been foud to correlate directly with stress levels. To check this enzyme, a sample of saliva is given.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term parturients

Exclusion Criteria:

* Diabetes
* Preterm labor
* Mouth pathologies

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Stress levels | 1 year

SECONDARY OUTCOMES:
hemodynamic parameters | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Orbach-Zinger, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tikvah, Israel